CLINICAL TRIAL: NCT01588951
Title: Consolidation Therapy for Acute Myeloid Leukemia Guided by Leukemia Stem Cell Behavior
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1227; NA_00071844 (Other: JHMIRB)
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Transplantation, Homologous; Bone Marrow Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No Leukemia Stem Cells - Consolidation (Experimental): Without LSC, standard cytarabine consolidation
  Interventions: Drug: Cytarabine consolidation
- Leukemia Stem Cells - Consolidation (Experimental): LSC present, randomized to cytarabine consolidation
  Interventions: Drug: Cytarabine consolidation
- Leukemia Stem Cells - Transplant (Experimental): LSC present, randomized to allogeneic transplant
  Interventions: Drug: Allogeneic transplant

INTERVENTIONS:
Drug: Cytarabine consolidation — Cytarabine-based consolidation per institutional standards.
  Other Names: HiDAC
  Arms: Leukemia Stem Cells - Consolidation; No Leukemia Stem Cells - Consolidation
Drug: Allogeneic transplant — Allogeneic stem cell transplant per institutional standards.
  Other Names: Bone marrow transplant; Stem cell transplant; Hematopoietic stem cell transplant; BMT; HSCT
  Arms: Leukemia Stem Cells - Transplant

SUMMARY:
The primary objective of the trial is to compare the two-year relapse-free survival (RFS) of patients with acute myeloid leukemia (AML), presumed to be at high risk for relapse due to the presence of leukemia stem cells (LSCs) in their bone marrow at first complete remission (CR1), who receive either standard cytarabine-based chemotherapy or allogeneic stem cell transplantation (SCT).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Able to give informed consent
3. New diagnosis of AML, other than APL or poor-risk AML, as defined in section 3.2

Exclusion criteria:

1. Has already had a bone marrow biopsy and aspirate to assess remission status after induction therapy
2. Any debilitating medical or psychiatric illness that would preclude ability to give informed consent or receive optimal treatment and follow-up
3. Pregnancy: Women of childbearing potential who are β- HCG+

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Showel, MD, Study Chair — JHU
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Transplant
Started | 2 | 2 | 6
Completed | 2 | 2 | 5
Not Completed | 0 | 0 | 1
Not completed — Ineligible in retrospect | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Transplant | Total
Number analyzed (Participants) | 2 | 2 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 6
  >=65 years | 0 | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 0 | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 0 | 2 | 4 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Description: Percentage of participants alive and without relapsed disease at two years.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | No Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Transplant
Number analyzed (Participants) | 2 | 2 | 5
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Collected monthly for up to 3.5 years.
Description: Only unexpected adverse events, grades III-IV acute GVHD, and chronic GVHD were collected.
Arm/Group | No Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Consolidation | Leukemia Stem Cells - Transplant
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT01588951/Prot_SAP_000.pdf